CLINICAL TRIAL: NCT01741194
Title: A 26-Week, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Investigate the Effects of Daily Administration of AC-1204 in Participants With Mild to Moderate Alzheimer's Disease (AD) With an Optional 26-Week Open Label Extension
Brief Title: AC-1204 26-Week Long Term Efficacy Response Trial With Optional Open-label Ext
Acronym: NOURISH-AD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AC-12-010
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AC-1204 (Experimental): Powder formulation (40 g) mixed with 4-8 ounces of water, other liquid or soft food as preferred, and shaken or blended until fully mixed. Each dosing unit of AC-1204 contains 20 g of the active ingredient, caprylic triglyceride.
  Interventions: Drug: AC-1204
- Placebo (Placebo Comparator): Placebo is an isocaloric formulation prepared to be virtually identical to AC-1204 in appearance, odor and taste. Powdered formulation is mixed with 4-8 ounces of water, other liquid or soft food as preferred, and shaken or blended until fully mixed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AC-1204 — AC-1204 taken once daily, by mouth
  Arms: AC-1204
Drug: Placebo — Placebo taken once daily, by mouth
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of daily dosing of AC-1204 on cognition, activities of daily living, resource utilization, quality of life, pharmacokinetic measures and safety among participants with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Dementia status of mild to moderate
* CT or MRI scan within 18 months prior to screening compatible with a diagnosis of probable Alzheimer's disease
* Score on the Wechsler Memory Scale - Logical Memory II recall below a pre-determined cut-off, adjusted for education level
* Confirmed apolipoprotein E genotype prior to randomization
* Prior and current use of medication that corresponds with protocol requirements
* Stable medical condition, with the exception of dementia, for at least 3 consecutive months prior to screening
* No active suicidal thoughts within 6 months of screening, no active history of suicide attempt in the previous 2 years, no more than 1 lifetime suicide attempt, no serious suicidal risk
* Able to comply with protocol testing and procedures for the duration of the study
* Has a permanent caregiver (caregiver is not expected to change during the course of the study) who is willing to attend all visits, oversee the participant's compliance with protocol procedures and study medication administration, and report on the participant's status
* Resides in the community (includes assisted living facilities, but excludes long-term care nursing facilities)
* Both participant and caregiver have the ability to read and write in English or Spanish and have hearing, vision and physical abilities adequate to perform the assessments (corrective aids allowed)
* Participant and caregiver have provided full written informed consent prior to the performance of any protocol-specified procedure. If participant is unable to provide informed consent due to cognitive status, provision of informed consent by cognitively intact legally acceptable representative (where this is in accordance with local laws, regulations and ethics committee policy)
* Participant is able to ingest oral medication

Exclusion Criteria:

* Current use, or use within 3 months of baseline, of medium-chain triglyceride-containing products
* Use of any other investigational agent within 60 days prior to screening
* Known allergy or hypersensitivity to milk or soy products
* In the opinion of the investigator, presence or history of advanced, severe, progressive or unstable disease of any type that could interfere with protocol assessments or put the participant at particular risk
* Any medical or neurological condition other than Alzheimer's disease that could explain the patient's dementia
* History or clinical laboratory evidence of moderate congestive heart failure
* Clinically significant ECG abnormalities at screening
* History of new cardiovascular events within 6 months prior to baseline
* History of or current psychiatric illness
* Major depression as determined by Cornell Scale for Depression in Dementia
* Insulin-dependent diabetics
* Systolic blood pressure > 165 mmHg or diastolic blood pressure > 95 mmHg
* Drop of 20 mm Hg systolic blood pressure or greater upon standing upright from a seated position within 3 minutes at screening
* Clinically significant anemia at screening
* Clinically significant renal disease or insufficiency at screening
* Laboratory values for liver function tests > 2.5 times the upper limit of normal at screening or history of severe liver disease
* Fasting triglycerides > 2.5 times the upper limit of normal at screening
* Clinically significant B12 deficiency within 12 month prior to screening
* Inflammatory bowel disease or peptic ulcer disease.
* Participants with current or a history of (within the last 5 years) complicated reflux disease or severe GERD that is not well-controlled by medication.
* Irritable bowel syndrome, diverticular disease (e.g., diverticulosis or diverticulitis), or chronic gastritis (exclusionary if there has been a diagnosis or an acute event within 5 years prior to Screening.)
* Has donated ≥ 2 units of blood within the 2 months prior to screening
* History of alcohol or drug abuse within 6 months prior to screening, or positive urine drug test at screening
* Participant or caregiver is an immediate family member or employee of the clinical site, sponsor or sponsor's agents
* An alternative cause for dementia other than Alzheimer's disease as determined by a required CT or MRI scan within 18 months prior to screening
* History of neoplasm or malignancies within 5 years prior to screening, except for basal cell or squamous cell carcinoma of the skin
* Clinically significant hypothyroidism as determined thyroid function testing at screening
* Participant has scheduled or expected hospitalization and/or surgery during the course of the study

Ages: 66 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 418 (Actual)
Dates: Start 2013-03; Primary Completion 2016-10-24 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) | 26 weeks
  APOE(-) participants

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) | 8 and 17 weeks
  APOE(-) participants
Clock Draw Interpretation Scale (CDIS) | 8 and 17 weeks
  APOE(-) participants
Alzheimer's Disease Co-operative Study - Clinical Global Impression of Change (ADCS-CGIC) | 26 weeks
  APOE(-) participants
Alzheimer's Disease Co-operative Study - Activities of Daily Living (ADCS-ADL) | 26 weeks
  APOE(-) participants
Quality of Life - Alzheimer's Disease (QoL-AD) | 26 weeks
  APOE(-) participants
Resource Utilization in Dementia (RUD-Lite) | 26 weeks
  APOE(-) participants
Incidence of treatment-emergent adverse events | 26 weeks
  All participants

OTHER OUTCOMES:
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) | 26 weeks
  APOE(+) participants
Clock Draw Interpretation Scale (CDIS) | 26 weeks
  APOE(+) participants
Alzheimer's Disease Co-operative Study - Clinical Global Impression of Change (ADCS-CGIC) | 26 weeks
  APOE(+) participants
Alzheimer's Disease Co-operative Study - Activities of Daily Living (ADCS-ADL) | 26 weeks
  APOE(+) participants
Quality of Life - Alzheimer's Disease (QoL- AD) | 26 weeks
  APOE(+) participants
Resource Utilization in Dementia (RUD-Lite) | 26 weeks
  APOE(+) participants
Mini Mental State Exam (MMSE) | 26 weeks
  APOE(+) participants
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) | 52 weeks
  All participants
Alzheimer's Disease Co-operative Study - Clinical Global Impression of Change (ADCS-CGIC) | 52 weeks
  All participants
Alzheimer's Disease Co-operative Study - Activities of Daily Living (ADCS-ADL) | 52 weeks
  All participants
Quality of Life - Alzheimer's Disease (QoL - AD) | 52 weeks
  All participants
Resource Utilization in Dementia (RUD-Lite) | 52 weeks
  All participants
Clock Draw Interpretation Scale (CDIS) | 52 weeks
  All participants
Ketone body levels (BHB) | baseline, 8, 17 and 26 weeks
  All participants
Incidence of treatment-emergent adverse events | 52 weeks
  All participants
Mini Mental State Exam (MMSE) | 52 weeks
  All participants

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T Henderson, PhD, Study Director — Cerecin
Locations (82):
- United States (82):
  - University of Alabama at Birmingham, Department of Neurology, Memory Disorders Division, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Principals Research Group, Hot Springs, Arkansas
  - Clinical Trials, Inc., Little Rock, Arkansas
  - CITrials, Inc., Bellflower, California
  - Southern Research LLC, Beverly Hills, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Diligent Clinical Trials, Downey, California
  - UCSD Comprehensive Alzheimer's Program, La Jolla, California
  - Alliance Research Centers, Laguna Hills, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Collaborative Neuroscience Network, Long Beach, California
  - Alliance for Research, Long Beach, California
  - Renew Behavioral Health, Long Beach, California
  - Pacific Research Network, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Research Across America, Santa Ana, California
  - Neurological Research Institute, Santa Monica, California
  - Redwood Research Medical Group, Santa Rosa, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - IMMUNOe Research Centers, Centennial, Colorado
  - The Mile High Research Center, Denver, Colorado
  - Chase Medical Research of Greater New Haven, Hamden, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Meridian Research, Brooksville, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - The Roskamp Institute, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - NeuroTrials Research, Inc, Atlanta, Georgia
  - IU Health Partners Adult Neurology Clinic, Indianapolis, Indiana
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Alzheimers Disease Center, Quincy Medical Center, Somerville, Massachusetts
  - Springfield Neurology Associates, Springfield, Massachusetts
  - Borgess Research Institute, Kalamazoo, Michigan
  - Saint Louis University Medical School /Department of Neurology & Psychiatry, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - NeuroCognitive Institute, Mount Arlington, New Jersey
  - Alzheimer's Research Corporation, Paterson, New Jersey
  - The Cognitive Research Center of New Jersey, Springfield, New Jersey
  - Memory Enhancement Center of NJ, Toms River, New Jersey
  - Neurology Specialists of Monmouth County, West Long Branch, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - The Litwin-Zucker Research Center, Manhasset, New York
  - Parker Jewish Institute For Health Care & Rehabilitation, New Hyde Park, New York
  - NYU Langone Medical Center Comprehensive Center on Brain Aging, New York, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - Nathan S. Kline Institute Geriatric Psychiatry Program, Orangeburg, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Ani Neurology, PLLC dba Alzheimer's Memory Ctr, Charlotte, North Carolina
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Valley Medical Research, Centerville, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Insight Clinical Trials LLC, Shaker Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Drexel Neurological Associates, Philadelphia, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Clinical Research Solutions, Franklin, Tennessee
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Senior Adults Specialty Research, Inc, Austin, Texas
  - Texas Neurology, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
  - VA Puget Sound-Alzhemier's Disease Research Center, Seattle, Washington

REFERENCES:
- [Derived] Henderson ST, Morimoto BH, Cummings JL, Farlow MR, Walker J. A Placebo-Controlled, Parallel-Group, Randomized Clinical Trial of AC-1204 in Mild-to-Moderate Alzheimer's Disease. J Alzheimers Dis. 2020;75(2):547-557. doi: 10.3233/JAD-191302. PMID 32310169